CLINICAL TRIAL: NCT03387215
Title: Randomized, Double-Blind, Placebo-Controlled, Safety and Tolerability Study of Escalating Single Doses of ITI-214 in Patients With Systolic Heart Failure
Brief Title: Randomized, Double-Blind, Placebo-Controlled, Safety and Tolerability Study of ITI-214 in Patients With Heart Failure
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Intra-Cellular Therapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ITI-214-104
Record Dates: First submitted 2017-12-18; First posted 2018-01-02 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Heart Failure, Systolic
MeSH Terms: conditions — Heart Failure, Systolic | interventions — ITI-214

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 10 mg ITI-214 (Experimental): Single oral dose
  Interventions: Drug: ITI-214
- 30 mg ITI-214 (Experimental): Single oral dose
  Interventions: Drug: ITI-214
- 75 mg - 150 mg ITI-214 (Experimental): Single oral dose
  Interventions: Drug: ITI-214
- Placebo (Placebo Comparator): Single oral dose
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ITI-214 — Oral
  Arms: 10 mg ITI-214; 30 mg ITI-214; 75 mg - 150 mg ITI-214
Other: Placebo — Oral
  Arms: Placebo

SUMMARY:
This is a Phase I/II randomized, double-blind, placebo-controlled, single rising dose study in patients with systolic heart failure to evaluate the safety and tolerability of ITI-214.

ELIGIBILITY:
Inclusion Criteria:

* NYHA class II-III heart failure
* Ejection fraction equal to or below 35%
* On stable heart failure drug treatment

Exclusion Criteria:

* Considered medically inappropriate for study participation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

PRIMARY OUTCOMES:
Echocardiogram with Doppler imaging and hemodynamic monitoring | 2 hours
  Cardiac systolic and diastolic function

SECONDARY OUTCOMES:
12-lead electrocardiogram (ECG) | 2 hours
  Safety and tolerability
Hemodynamic monitoring | 5-6 hours
  Cardiac systolic and diastolic function
Number of patients with treatment-emergent adverse events | 5 days
  Safety and tolerability

OTHER OUTCOMES:
Plasma and urine levels of cAMP and cGMP as Exploratory biomarkers | 2 hours
  Pharmacodynamics

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Johns Hopkins University, Baltimore, Maryland
  - Duke Clinical Research Institute, Durham, North Carolina

REFERENCES:
- [Derived] Gilotra NA, DeVore AD, Povsic TJ, Hays AG, Hahn VS, Agunbiade TA, DeLong A, Satlin A, Chen R, Davis R, Kass DA. Acute Hemodynamic Effects and Tolerability of Phosphodiesterase-1 Inhibition With ITI-214 in Human Systolic Heart Failure. Circ Heart Fail. 2021 Sep;14(9):e008236. doi: 10.1161/CIRCHEARTFAILURE.120.008236. Epub 2021 Aug 31. PMID 34461742